CLINICAL TRIAL: NCT06045897
Title: Determination of EEG Microstates Associated With Mental Disorders in At-Risk States (Détermination Des Microétats EEG associés Aux Troubles Psychiques Dans Les États à Risque - DEMETER)
Brief Title: EEG Microstates Across At-Risk Mental States
Acronym: DEMETER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A01919-32
Record Dates: First submitted 2021-07-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Psychotic Disorders; Autism Spectrum Disorder; Major Depressive Disorder; Schizophrenia
Keywords: electroencephalography; at risk mental state; ultra high risk; first episode psychosis; schizophrenia; autism spectrum disorder; EEG microstates; polysomnography; sensorimotor integration; prosody; hypnosis
MeSH Terms: conditions — Psychotic Disorders; Autism Spectrum Disorder; Depressive Disorder, Major; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Major depressive disorder (Experimental): Major depressive disorder as defined by DSM-5 classification
  Interventions: Device: EEG 64 channels; Device: Polysomnography 19 electrodes; Biological: Biological sampling; Device: Voice recording
- Autism spectrum disorder (Experimental): Autism spectrum disorder as defined by DSM-5 classification
  Interventions: Device: EEG 64 channels; Device: Polysomnography 19 electrodes; Biological: Biological sampling; Device: Voice recording
- At risk mental state (Experimental): At risk mental state as defined in the CAARMS
  Interventions: Device: EEG 64 channels; Device: Polysomnography 19 electrodes; Biological: Biological sampling; Behavioral: Virtual reality; Device: Voice recording
- First episode psychosis (Experimental): Any DSM-5 category associated with psychotic symptoms
  Interventions: Device: EEG 64 channels; Device: Polysomnography 19 electrodes; Biological: Biological sampling; Behavioral: Virtual reality; Device: Voice recording
- Schizophrenia (Experimental): Schizophrenia as defined by DSM-5 classification
  Interventions: Device: EEG 64 channels; Device: Polysomnography 19 electrodes; Biological: Biological sampling; Device: Voice recording
- Healthy controls (Experimental): Healthy controls with no history of neurodevelopmental disorder or psychotic disorder in a first degree relative
  Interventions: Device: EEG 64 channels; Device: Polysomnography 19 electrodes; Behavioral: Light hypnosis; Biological: Biological sampling; Behavioral: Virtual reality; Device: Voice recording

INTERVENTIONS:
Device: EEG 64 channels — 64-channel EEG in wake and resting conditions for 1h30, with oculogram, electromyogram and electromyogram and electrocardiogram. Five minutes of eyes closed will be used for microstate analysis. 1h30 will be used for the sensorimotor task.
Device: Polysomnography 19 electrodes — Overnight polysomnography with 19 EEG channels and ventilatory polygraphy.
Behavioral: Light hypnosis — Healthy controls will undergo a 5 min light hypnosis exercise that will be focused on proprioception.
  Arms: Healthy controls
Biological: Biological sampling — Blood samples will be taken for genetic, epigenetic, proteomic, and metabolomic studies.
Behavioral: Virtual reality — Participants will undergo a virtual reality task using a head-mounted display, and their multidimensional self will be assessed prior to and after the task via the self-reference effect on episodic memory.
  Arms: At risk mental state; First episode psychosis; Healthy controls
Device: Voice recording — A double channel audio recorder will be used during 30 min to assess voice characteristics of all subjects.

SUMMARY:
The goal of this observational study is to compare subjects with at-risk-mental-state, early psychosis, schizophrenia, depression, and autism spectrum disorders, with healthy controls (N = 21 x 6). The main questions it aims to answer are:

* are EEG microstate anomalies associated with diagnosis, clinical and functional prognosis, both in resting conditions and during sleep ?
* are EEG microstates anomalies associated with differences in sensorimotor integration, prosodic and conversational, interoceptive, and narrative self ?
* an ancillary study will be to see whether in healthy controls EEG microstate properties vary under light hypnosis conditions.

Participants will:

* undergo deep phenotyping based on psychopathology and neuropsychological assessments
* undergo a high-resolution EEG (64 electrodes) with a resting period and a sensorimotor task; and healthy controls will have a light hypnosis period.
* undergo a recording of the characteristics of their voice (tone, prosody)
* undergo a one-night polysomnography
* undergo MRI and biological sampling for multi-omic analyses
* undergo a virtual reality experience

DETAILED DESCRIPTION:
* Aim of the study: EEG microstates translate the resting-state temporal dynamics of neuronal networks throughout the brain. Here, the investigators aim to see whether EEG microstate anomalies could constitute markers of psychiatric disorders.
* Methods: six groups of 21 participants each will be included. There will be five groups of participants with psychiatric disorders (at-risk-mental state - ARMS, first-episode psychosis - FEP, schizophrenia - SCZ, major depressive disorder - MDD, and autism spectrum disorders - ASD) and one group of healthy controls. Our main objective is to test differences in means between the groups, at rest and during sleep, for each of the variables characterizing each of the microstates (duration, frequency, occupation time) as well as, secondarily, EEG measures of connectivity (somatosensory evoked potentials), cortical excitability (alpha-band power), and prosodic and conversational linguistic measures.

  * Regarding the microstates measures: a five minute eyes-closed resting-state EEG with 64 channels will be recorded (as part of the larger task including the sensorimotor task described below). A minimal preprocessing will be done with the MNE EEG software on Python, which includes a bandpass filter between 0.5 and 40 Hz, rereferencing to the mean, and visual and automatic correction for artifacts. Each recording will be visually reanalyzed by clinical neurophysiologists to ensure it is indeed an alpha-dominant, resting rhythm without any residual artifact. Microstate analysis will be done using the Pycrostates package. Global field power (GFP) will be determined for each participant. Only EEG topographies at GFP peaks will be retained to determine microstates' topographies, through a modified K-means clustering. For each subject the same number of GFP peaks will be extracted and concatenated into a single data set for clustering. A combined score will be used to compute the optimal number of clusters. The resulting clusters will be backfitted to each individual maps. Temporal smoothing will be used to ensure that periods of inter-peak noise, of low GFP, did not interrupt the sequences of quasi-stable segments. For each subject, three parameters will be computed for each microstate class: frequency of occurrence ("occurrence"), temporal coverage ("coverage") and mean duration. Occurrence is the average number of times a given microstate occurs per second. Coverage (in %) is the percentage of total analysis time spent in a given microstate. Mean duration (in ms) is the average time during which a given microstate was present in an uninterrupted manner (after temporal smoothing).
  * Regarding the linguistic measures: each participant undergoes a semi-structured interview with a trained experimenter. Both the participant and the interviewer wear head-set AKG-C544L condenser microphones, connected via AKG MPA VL phantom adaptors to a Zoom H4n Pro Handy recorder. Speech is digitally recorded at a sampling rating of 44000 Hz (16-bit). The distance between the mouth and the microphone is kept as constant as possible (2 cm) to assure consistent levels of vocal loudness. The interviews are done in a quiet room to limit environmental noise; the two interactants are placed as far as possible, to prevent crosstalk (i.e. speech of the interviewer caught by participant's microphone and vice versa). The .wav files obtained from the recordings are annotated using the Praat software and subsequently analysed with Praat and R. Prosodic features are extracted using the Prosogram tool (a set of Praat scripts, open-source) and a new modified version of scripts from the Prosogram tool. Turn-taking variables are extracted with new combined Praat and R scripts.
  * Regarding the sensorimotor intergration measures: the sensorimotor integration is investigated using a visuo-haptic task. On each trial, the participant, seated in front of a screen, has a visual instruction (a point to the right or left of the screen). The task consists of pressing one of the two buttons positioned on each side of the body with the index finger of the corresponding hand according to the visual instruction. A vibrotactile stimulator (small speakers wired to an Arduino electronic card modulated by an amplifier) is applied to the first dorsal interosseous muscle of both hands. 400 msec before the visual instruction, one of the two hands receives a tactile cue (vibration) on one hand for 100 msec. This cue is more or less reliable depending on the block. In some blocks, it is quite reliable, since 90% of the trials present the vibration and visual instruction congruently (indicating the same hand). Another condition is composed of only 50% of the congruent trials, and in this case, the tactile cue is not reliable. Two blocks with 70% congruent cases are carried out intermediately. Finally, a baseline block which does not contain any tactile cues is presented at the beginning and the end of the task. The order of the 90% and 50% blocks is randomized. The tactile and visual stimuli are generated with a MATLAB script. Each block consists of 100 trials, in total 500 trials. Electroencephalographic (EEG) data is recorded throughout the task, using a 64-channel EEG cap (from Biosemi) in order to record the electrical brain activity. The setup is coupled to an eyetracker, to control that the participant is fixating the cross at the center of the screen during each block.
  * Regarding the multidimensional self and episodic memory task (task design: Laboratoire Mémoire, Cerveau et Cognition): at baseline, participants will be submitted to self-reported questionnaires assessing their sense of minimal Self on 8 domains (Multidimensional Assessment of Interoceptive Awareness - Version 2) and sense of narrative Self on 5 domains (Tennessee Self Concept Scale - Short Form, Present). They will undergo a neuropsychological test assessing their visual episodic memory performance (Family Pictures from Wechsler Memory Scale-III). They will rate their current emotional state on a visual analogue scale on 4 domains (Mood Visual Analogue Scale). Following each of the two navigation sessions in virtual reality, which consist in a walk through a virtual city where participants encounter daily life events that aim to be incidentally encoded in episodic memory, associated with different levels of self-reference, participants will be submitted to self-reported questionnaires assessing their sense of embodiment on 4 domains (Embodiment Questionnaire), their sense of presence on 4 domains (Igroup Presence Questionnaire), and their cybersickness on 2 domains (Simulator Sickness Questionnaire). They will rate again their current emotional state on a visual analogue scale (Mood Visual Analogue Scale). Finally, participants will undergo two episodic memory tests: a free recall task and a recognition task. The free recall will be based on a verbal interview of 20 minutes, during which participants will be asked to recall all the events that they remember encountering in the virtual city. For each event, they will be asked to recall systematically and the most precisely possible: what was the event, where and when it happened during the navigation, in which of the two navigation it happened (source), who was the referent according to which the personal significance of the event was assessed, objective (perceptive) and subjective (phenomenological) details of the event, and if the event was vividly relived or felt merely familiar (Remember/Know procedure). The recognition test will be performed on a computer and programmed using the Python module Neuropsydia. All 32 encountered events mixed with 16 lures which were not encountered will be displayed successfully in a random order on a computer screen. For each event, several questions will be asked successfully and participants will click on what they consider the correct answer among several propositions: did they encounter the event (Yes/No), and if yes where it happened (among several possible localisations on a picture of the zone where the event occurred), when it happened (replacing the event in the chronological order with two other events), in which navigation (first or second navigation), and who was the referent (Me/Other). For each event, participants will also rate on scales ranging from 0 to 100: the degree of reliving or familiarity of the event (100 = Remember, 0 = Know), the perspective of the memory (100 = first-person perspective, 0 = third-person perspective), its vivacity, fidelity, emotional intensity, strength of associated bodily sensations, episodic self-reference, and semantic self-reference.

For all variables, the investigators will apply a repeated measures ANOVA, and use the following contrasts:

1. "ARMS, FEP, SCZ, ASD, MDD" vs. "Healthy subjects" (microstates are tested as markers of general psychopathology);
2. "ARMS, FEP, SCZ" vs "ASD, MDD" (microstates are tested as specific markers of psychosis; equivalently, the specificity of this signature for depression and ASD will be tested)
3. "ARMS" vs. "FEP" vs. "SCZ" (microstates are tested as evolutionary markers);
4. Finally, depending on the rate of transition to psychosis among UHRs, a comparison of "UHR-T" vs "UHR-NT" can be made (microstates are tested as predictive markers of psychosis All subjects will undergo a deep phenotyping including neuropsychology, psychopathology, neurological soft signs scales, as well as structural MRI, and genetic and epigenetic measures.

   * Hypothesis: imbalances in EEG microstates C and D are expected to be more pronounced across the spectrum of psychosis and in ASD compared to controls, MDD, and ARMS, and be associated with anomalies in somatosensory, interoceptive, and language characteristics.

ELIGIBILITY:
Inclusion Criteria:

* age between 15 and 30 years
* subjects meeting CAARMS criteria for stage Ia or Ib mental states at risk (for stage Ia, mild or nonspecific symptoms of psychosis or severe mood disorder, and mild functional impairment; for stage Ib, moderate symptoms below intervention threshold and moderate functional impairment)
* subjects meeting any DSM-5 criteria associated with a first onset of psychotic symptoms (first episode psychosis)
* subjects satisfying DSM-5 criteria for depressive disorder
* subjects meeting DSM-5 criteria for autism spectrum disorder
* healthy control subjects recruited from the general population

Exclusion Criteria:

* suicidal risk
* severe or non-stabilized somatic and neurological disorders
* epilepsy
* head trauma
* IQ below 70
* for healthy control subjects, a family history of psychosis is an exclusion criterion
* bipolar disorder
* obsessive-compulsive disorder
* substance use disorder, except for cannabis, tolerated up to 5 joints/day.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of EEG microstates | Three years
  Average number of times a given microstate occurs per second.
Coverage of EEG microstates | Three years
  Percentage of total analysis time spent in a given microstate.
Mean duration of EEG microstates | Three years
  Average time during which a given microstate was present in an uninterrupted manner (after temporal smoothing).

SECONDARY OUTCOMES:
Attention modulation | Three years
  Measurement of alpha band power (in Hz)
Cortical excitability and inhibition | Three years
  Measurement of mu and theta bands (in Hz)
Integration of sensory information: amplitudes | Three years
  Measurement of amplitudes (in µV) of somatosensory evoked potentials
Integration of sensory information: latencies | Three years
  Measurement of latencies (in msec) of somatosensory evoked potentials
Reaction time | Three years
  The adaptation of the reaction time (in msec) to the button press according to the probabilistic context of congruency is examined.
Speech rate | Three years
  Measurement of number of syllables/sec in the recording of the subjects
Fundamental frequency | Three years
  Measurement of the fundamental frequency (in Hz)
Pitch mean | Three years
  Measurement of the pitch mean (in semi-tones)
Pitch range | Three years
  Measurement of the pitch range (in semi-tones)
Pitch gliss | Three years
  Measurement of the proportion of syllables with large pitch movement (in percents)
Pitch rises | Three years
  Measurement of the proportion of syllables with pitch rise (in percents)
Pitch falls | Three years
  Measurement of the proportion of syllables with pitch fall (in percents)
Nuclei duration | Three years
  Sum of durations for syllable nuclei for the speaker (in seconds)
Internuclei Duration | Three years
  Sum of durations between successive nuclei for the speaker (in seconds)
Intrasyllabic Trajectory | Three years
  Pitch trajectory (sum of absolute intervals) within syllabic nuclei, divided by duration (in semitones per second)
Intersyllabic Trajectory | Three years
  Pitch trajectory (sum of absolute intervals) between syllabic nuclei (except pauses or speaker turns), divided by duration (in semitones per second)
Percentage of turns interviewer | Three years
  Interviewer's total number of turns divided by the total number of turns of the dialogue (in percents)
Percentage of turns participant | Three years
  Participant's total number of turns divided by the total number of turns of the dialogue (in percents)
Interviewer's Floor Occupation | Three years
  Portion of time where only the interviewer is speaking (in percents)
Participant's Floor Occupation | Three years
  Portion of time where only the participant is speaking (in percents)
Overlap | Three years
  Portion of time where both interactants are speaking (in percents)
Mutual silence | Three years
  Portion of time where both interactants are silent (in percents)
Between-Overlap | Three years
  Turn transition composed of overlapping speech from both interlocutors (in percents)
Gap | Three years
  Silent interval between turn transitions (in percents)
Within-Overlap | Three years
  Passages of overlapping speech not followed by a change of speaker (in percents)
Floor Transfer Offset | Three years
  Measures of gaps (positive values) and overlaps (negative values) in milliseconds
Interviewer's Speaking Turn Duration | Three years
  Average duration of interviewer's speaking turns in milliseconds
Interviewer's Silent Turn Duration | Three years
  Average duration of interviewer's pauses in milliseconds
Participant's Speaking Turn Duration | Three years
  Average duration of the participant's speaking turns in milliseconds
Participant's Silent Turn Duration | Three years
  Average duration of the participant's pauses in milliseconds
Minimal self | Three years
  Measure on the Multidimensional Assessment of Interoceptive Awareness - Version 2; Min = 0, max =185; Higher score is a better outcome
Narrative self | Three years
  Measure on the Tennessee Self Concept Scale - Short Form, Present; Min = 21, max = 105; Higher score is a better outcome
Visual episodic memory performance | Three years
  Measure on the Family Pictures from Wechsler Memory Scale-III (standardized score)
Current emotional state before the task | Three years
  Measure on the Mood Visual Analogue Scale; Min = 0, max = 100; Higher score is a better outcome
Embodiment | Three years
  Measure on the Embodiment Questionnaire; Min = -3, max = 3; Higher score is a better outcome
Presence | Three years
  Measure on the Igroup Presence Questionnaire; Min = -42, max = 42; Higher score is a better outcome
Cybersickness | Three years
  Measure on the Simulator Sickness Questionnaire; Min = 0, max = 48; Higher score is a worse outcome
Current emotional state after the task | Three years
  Measure on the Mood Visual Analogue Scale; Min = 0, max = 100; Higher score is a better outcome
Recognition task: "What" 1 | Three years
  Proportion of hits (number of recognised events divided by total number of events) (in percents)
Recognition task: "What" 2 | Three years
  Proportion of false alarms (number of falsely recognised lures divided by total number of lures) (in percents)
Recognition task: "What" 3 | Three years
  Hit mean reaction time (in seconds)
Recognition task: "What" 4 | Three years
  False alarm mean reaction time (in seconds)
Recognition task: "When" | Three years
  Proportion of correct "When" answers (number of correct "When" answers divided by number of hits) (in percents)
Recognition task: "Where" | Three years
  Proportion of correct "Where" answers (in percents)
Recognition task: "Source" | Three years
  Proportion of correct "Source" answers (in percents)
Recognition task: "Binding What-When-Where" | Three years
  Mean of (What + When + Where) (in percents)
Recognition task: "Binding What-When-Where-Source" | Three years
  Mean of (What + When + Where + Source) (in percents)
Recognition task: "Referent" | Three years
  Proportion of correct "Referent" answers (in percents)
Recognition task: "Remember/Know" | Three years
  Mean (a score between 0 and 100)
Recognition task: "Perspective" | Three years
  Mean (a score between 0 and 100)
Recognition task: "Vivacity" | Three years
  Mean (a score between 0 and 100)
Recognition task: "Fidelity" | Three years
  Mean (a score between 0 and 100)
Recognition task: "Emotional intensity" | Three years
  Mean (a score between 0 and 100)
Recognition task: "Strength of associated bodily sensations" | Three years
  Mean (a score between 0 and 100)
Recognition task: "Episodic self-reference" | Three years
  Mean (a score between 0 and 100)
Recognition task: "Semantic self-reference" | Three years
  Mean (a score between 0 and 100)
Free recall: "What" | Three years
  Proportion of recalled events (in percents)
Free recall: "When" | Three years
  Proportion of correct "When" answers (in percents)
Free recall: "Where" | Three years
  Proportion of correct "Where" answers (in percents)
Free recall: "Source" | Three years
  Proportion of correct "Source" answers (in percents)
Free recall: "Binding What-When-Where" | Three years
  Mean of (What + When + Where) (in percents)
Free recall: "Binding What-When-Where-Source" | Three years
  Mean of (What + When + Where + Source) (in percents)
Free recall: "Referent" | Three years
  Proportion of correct "Referent" answers (in percents)
Free recall: "Objective details" | Three years
  Mean number of objective details
Free recall: "Subjective details" | Three years
  Mean number of subjective details
Free recall: "Remember/Know" 1 | Three years
  Proportion of "Remember" answers (in percents)
Free recall: "Remember/Know" 2 | Three years
  Proportion of "Know" answers (in percents)

CONTACTS AND LOCATIONS:
Overall Officials: Anton Iftimovici, MD, PhD, Principal Investigator — GHU Paris Psychiatrie et Neurosciences
Locations (1):
- Centre de Recherche Clinique, Hôpital Sainte-Anne, GHU Paris Psychiatrie et Neurosciences, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iftimovici A, Marchi A, Ferat V, Pruvost-Robieux E, Guinard E, Morin V, Elandaloussi Y, D'Halluin A, Krebs MO, Chaumette B, Gavaret M. Electroencephalography microstates imbalance across the spectrum of early psychosis, autism, and mood disorders. Eur Psychiatry. 2023 May 29;66(1):e41. doi: 10.1192/j.eurpsy.2023.2414. PMID 37246142
- [Background] Gavaret M, Iftimovici A, Pruvost-Robieux E. EEG: Current relevance and promising quantitative analyses. Rev Neurol (Paris). 2023 Apr;179(4):352-360. doi: 10.1016/j.neurol.2022.12.008. Epub 2023 Mar 10. PMID 36907708
- [Derived] Lucarini V, Alouit A, Yeh D, Le Coq J, Savatte R, Charre M, Louveau C, Houamri MB, Penaud S, Gaston-Bellegarde A, Rio S, Drouet L, Elbaz M, Becchio J, Pourchet S, Pruvost-Robieux E, Marchi A, Moyal M, Lefebvre A, Chaumette B, Grice M, Lindberg PG, Dupin L, Piolino P, Lemogne C, Leger D, Gavaret M, Krebs MO, Iftimovici A. Neurophysiological explorations across the spectrum of psychosis, autism, and depression, during wakefulness and sleep: protocol of a prospective case-control transdiagnostic multimodal study (DEMETER). BMC Psychiatry. 2023 Nov 21;23(1):860. doi: 10.1186/s12888-023-05347-x. PMID 37990173